CLINICAL TRIAL: NCT01505478
Title: Comparing an Automated to a Conventional Sepsis Clinical Prediction Rule
Status: Withdrawn | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: New York University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven Horng, MD, Instructor in Emergency Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2011P000356
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2012-01

CONDITIONS: Sepsis
Keywords: Sepsis; Clinical Prediction Rule; Clinical Informatics; Machine Learning
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients admitted with infection: All consecutive ED patients during the study period that have been admitted and identified to have a suspected infection at ED disposition using a data collection tool

SUMMARY:
The investigators will conduct a prospective cohort study to compare an automated sepsis severity score to a conventional clinical prediction rule to risk stratify patients admitted from the emergency department (ED) with suspected infection for 28 day in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult (age 18 or older) Emergency Department (ED) patients during the study period that have been admitted from the ED and identified by the treating clinician to have a suspected infection at the time of ED disposition will comprise our study population.

Exclusion Criteria:

* No patients will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted from the Emergency Department with suspected infection.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07

PRIMARY OUTCOMES:
28 day in-hospital mortality
  The primary endpoint is the AUC of a model to predict 28 day all cause in-hospital mortality. Patients discharged or transferred to another hospital before 28 days will be assumed to be alive at 28 days.

SECONDARY OUTCOMES:
ICU Admission
  The secondary endpoint is ICU admission from the ED or within 24 hours from the floor.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Horng, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States